CLINICAL TRIAL: NCT06900439
Title: Exploring Glycemic Responses Through Continuous Monitoring in a Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zoe Global Limited (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZOE PREDICT REFINE
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Gut Microbiome; Glucose Control
Keywords: CGM; Continuous Glucose Monitor; Glucose; Gut Microbiome; Healthy Population; Glycemic Response
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: A single-arm mechanistic intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dietary Intervention (Experimental): Dietary intervention using a standardized test meal after which the postprandial glucose response is measured.
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — To carry out a dietary intervention using a standardized test meal where the participant's postprandial glucose to the meal is measured with a continuous glucose monitor and compared to the participant's postprandial glucose from the same standardized test meal 4 months prior.

SUMMARY:
PREDICT REFINE is a sub-study of PREDICT 3 with the primary aim of exploring glycemic responses through continuous glucose monitoring in a healthy population. The study will explore glycemic responses to a standardised test meal before and after a personalised dietary programme.

The sub-study will include wearing a Continuous Glucose Monitor for 14 days, collecting information around diet and health, providing a stool sample, and consuming a standardised test meal.

By conducting this study researchers hope to better understand Continuous Glucose Monitoring accuracy and variability in healthy individuals, the impact of diet on glycemic responses over time, and potential mechanisms by which changes in microbiome health may influence glycemic control.

DETAILED DESCRIPTION:
PREDICT REFINE is a single-arm mechanistic intervention study designed as a sub-study of PREDICT 3. The primary objective is to explore glycemic responses through continuous glucose monitoring (CGM) in a healthy population, specifically examining responses to a standardized test meal before and after a personalised dietary programme.

Study Population and Recruitment:

The study population consists of individuals who have previously enrolled in the commercial ZOE testing program, consented to participate in the PREDICT 3 study, and provided consent for scientific research at ZOE. Prospective participants will be selected based on predefined inclusion and exclusion criteria by the study management team. Recruitment will be conducted via email, with potential participants receiving a Participant Information Sheet. A minimum of 24 hours will be provided for individuals to consider participation. Those interested will complete an online screening form via a secure survey platform, and eligible participants will be asked to provide informed consent.

Study Design and Procedures:

Following informed consent, participants will undergo the following study tasks in a 14 day timeframe:

1. Continuous Glucose Monitoring: Participants will wear a CGM device for 14 days to record continuous data on blood glucose responses.
2. Data Collection: Participants will be required to provide comprehensive information about their diet and health during the study period. This will include completing food logs, a food frequency questionnaire, and a health + lifestyle questionnaire on a mobile app.
3. Biological Sample Collection: Participants will provide a stool sample, which will be analyzed using metagenomic sequencing.
4. Consume a Standardized Test Meal: Participants will consume a standardized test meal under controlled conditions.

As participants will be recruited from the PREDICT 3 study, the above tasks would have been completed at baseline, ~4 months prior to the start of the sub study while participating in PREDICT 3. Study consent will allow baseline and endpoint data (collected as part of this sub-study) to be connected.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the ZOE product & purchased a Gut Health Retest at month 4
* Any sex
* Minimum 18 years of age
* Body mass index (BMI) greater than or equal to 18.5 kg/m2
* If under care for any chronic medical conditions (including type 2 diabetes), you have confirmed with your treating physician that this sub study is safe for you. This does not apply to conditions listed in the exclusion criteria.
* Able and willing to comply with the study protocol and provide informed consent before your ZOE Gut Health Retest is fulfilled and posted.
* Live in the United Kingdom

Exclusion Criteria:

* Cannot safely eat the standardised meals (part of the ZOE product) which contain standard UK ingredients, e.g. due to allergy or recent gastrointestinal surgery
* Cannot safely use the cgm (per manufacturer's contraindications for use including critically ill, pregnant, receiving dialysis, or have an implantable medical device)
* Are pregnant
* Have had a heart attack (myocardial infarction), stroke/transient ischemic attack (TIA), or major surgery in the last two months
* Are unable to read and write in English, as the ZOE app is only available in English.
* Are diagnosed with type 1 diabetes and/or require the use of exogenous insulin or oral hypoglycaemic medications to regulate blood sugar levels
* Have an active eating disorder (e.g. anorexia nervosa or bulimia nervosa)
* Have an active gut or digestive system disease (e.g. IBD, Crohn's disease or ulcerative colitis)
* Are undergoing chemotherapy treatment for cancer
* Unable to complete study tasks by 31 May 2025

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1189 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Glycaemic Control | Baseline and Month 4
  Measurement of glycaemic control with a continuous glucose monitor (CGM).

SECONDARY OUTCOMES:
Gut Microbiome Composition | Baseline and Month 4
  The measurement of relative abundance of microbiome species, derived from metagenomic analysis of stool samples.
Gut Microbiome Diversity | Baseline and Month 4
  The measurement of diversity metrics (e.g. richness, evenness, ranking of species associated with diet and health) derived from metagenomic analysis of stool samples.

OTHER OUTCOMES:
Dietary Intake | Baseline and Month 4
  The measurement of habitual and acute dietary intake through a food frequency questionnaire and food logs.

CONTACTS AND LOCATIONS:
Locations (1):
- ZOE Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No